CLINICAL TRIAL: NCT04276519
Title: Randomized Controlled Trial to Investigate the Feasibility of a New Protocol for Treatment of Acute Low Back Pain and Sciatica From Lumbar Radiculopathy and Intervertebral Disc Herniation: Non-invasive Position-Induced Opening of the Intervertebral Foramen
Brief Title: Position-Induced Opening of the Intervertebral Foramen is Efficient to Treat an Acute Lumbosacral Radiculopathy Caused by Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital Sveti Duh (Other)
Responsible Party: Principal Investigator, Sinisa Poznic, Master of Science in Physiotherapy, General Hospital Sveti Duh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01-2748
Record Dates: First submitted 2020-02-10; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Radiculopathy Lumbar; Disk Herniated Lumbar; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Experimental group and a control group. Prospective, randomised, clinical study.
Who Masked: Participant
Masking Description: Participants didn't know in which group they were allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Physiotherapeutic non-invasive position-induced opening of the intervertebral foramen and pharmacological treatment with steroid antiinflammatory drugs - dexamethasone, nonsteroid antiinflammatory drugs and pain killers - tramadol.
  Interventions: Procedure: Physiotherapeutic, non-invasive position-induced opening of the intervertebral foramen
- Control group (Active Comparator): Pharmacological treatment with steroid antiinflammatory drugs - dexamethasone, nonsteroid antiinflammatory drugs and pain killers - tramadol.
  Interventions: Procedure: Physiotherapeutic, non-invasive position-induced opening of the intervertebral foramen

INTERVENTIONS:
Procedure: Physiotherapeutic, non-invasive position-induced opening of the intervertebral foramen — Opening of the mechanical interface of the nerve root, neurodynamics

SUMMARY:
Efficiency of the conservative mechanical lumbosacral nerve root decompression, as an adjunct to pharmacological treatment, in the case of acute lumbosacral radiculopathy.

DETAILED DESCRIPTION:
Non-invasive Position-Induced Opening of the Intervertebral Foramen in sidelying position, as an adjunct to pharmacological treatment, was used in the case of acute lumbosacral radiculopathy.

20 examinees were split into two groups, 10 in the experimental and 10 in the control group. Experimental group was given positional opening of the intervert. foramen, together with pharmacological treatment - steroid antiinflammatory drug - dexamethasone, nonsteroid antiinflammatory drugs and pain killers while control group was given just the same pharmacological treatment and recommended rest.

Measured dependent variables were:

1. Visual analogue pain scale (VAS) for the low back and radiculopathy, separately
2. Straight leg raise in supine position - nerve mobility test
3. EuroQol questionnaire - general health condition questionnaire
4. Oswestry questionnaire - activities of daily living (ADL) specific questionnaire for low back pain and lumbosacral radiculopathies Inclusive criteria were: Age between 20 - 60, lumbar disc herniation recognized by the MRI, lumbosacral radiculopathy with symptoms such as radicular pain, sensation dysfunctions or motor dysfunctions, recognized by electromyography (EMG) diagnostics.

Exclusive criteria: age more than 60, degenerative lumbar stenosis, spondylolisthesis, vertebra fractures, tumours.

Conclusion: Physiotherapy with a positional, mechanical decompression of the compressed lumbosacral nerve root, as an adjunct to pharmacological treatment, is proved to be efficient with the lumbosacral radiculopathy. It is recommended to be applied since the first day of a patient admittance in the hospital if there is a position that can reduce the pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 - 60
2. Lumbar disc herniation proved by MRI
3. Lumbosacral radiculopathy with symptoms of radicular pain, sensation dysfunction, and motor dysfunction proved by EMG diagnostics.

Exclusion Criteria:

1. Age older than 60
2. Degenerative lumbar stenosis
3. Spondylolisthesis
4. Vertebrae fractures
5. Tumor metastasis

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain scale for low back pain (LBP) Visual analogue scale for radiculopathy | Change from baseline pain subjectively reported value by Visual Analogic Scale compared to same values at discharge (mean value 8 days)
  Pain descriptor
Straight leg raise | Change from baseline nerve mobility objectively reported value by straight leg raise compared to same values at discharge (mean value 8 days)
  Nerve mobility test for lower lumbar nerve roots and n. ischiadicus
EuroQol questionnaire | Change from baseline general health condition subjectively reported value by EuroQol questionnaire compared to same values at discharge (mean value 8 days)
  General health condition questionnaire
Oswestry questionnaire | Change from baseline activity of daily living specific questionnaire for low back pain and lumbosacral radiculopathy subjectively reported value by Oswestry questionnaire compared to same values at discharge (mean value 8 days)
  ADLs specific questionnaire for LBP and lumbosacral radiculopathy

CONTACTS AND LOCATIONS:
Overall Officials: Anita Marcinko Budincevic, Study Chair — Clinic of Neurology, Sveti Duh Clinical Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Holy Spirit Clinical Hospital — http://www.kbsd.hr/
- See also: Clinical neurodynamics — http://www.neurodynamicsolutions.com/